CLINICAL TRIAL: NCT02921438
Title: A Prospective Multi-centre Observational Study to Evaluate the Diagnostic Accuracy of a Portable Magnetocardiograph Device for Acute Coronary Syndrome (ACS), Focusing on Rule-out Capability, in Patients Who Present to the Emergency Department With Chest Pain Symptoms Consistent With ACS.
Brief Title: VitalScan MCG Rule-out Multi-centre Pivotal Study - UK
Acronym: MAGNET-ACS
Status: Completed | Type: Observational
Sponsor: Creavo Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP 003
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2018-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; NSTE ACS; NSTEMI; Unstable Angina Pectoris; Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Cardiovascular Diseases; Heart Diseases; Myocardial Ischemia; Non-ST Elevated Myocardial Infarction; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain patients presenting to the ED: All patients that present to the emergency department with chest pain and potentially other symptoms consistent with ACS and meet all eligibility criteria will undergo VitalScan Magnetocardiograph.
  Interventions: Device: VitalScan Magnetocardiograph

INTERVENTIONS:
Device: VitalScan Magnetocardiograph — A passive, non-contact, mobile medical device that measures, displays, stores, and retrieves magnetic fluctuations caused by heart activity at a patient's bedside.

SUMMARY:
The study is a prospective multi-centre observational study to evaluate a portable magnetocardiograph device for the rule-out of acute coronary syndrome (ACS) in patients who present to the emergency department with chest pain and other symptoms consistent with ACS.

DETAILED DESCRIPTION:
Few, if any, studies have evaluated the rule-out (R/O) of non-ST-segment elevation (NSTE) ACS which requires the sensitivity and negative predictive value (NPV) of the test to approach 100%. An alternative triage approach, utilizing a portable magnetocardiography (MCG) instrument in the emergency setting, may lead to a more accurate R/O for NSTEMI, UA, and clinically significant non-ACS coronary artery disease (CAD), in patients presenting to the ED with chest pain. MCG in the emergency setting is a new use of this non-invasive technique and may serve as an adjunctive aid that can improve cardiac triage for NSTE ACS and clinically significant CAD.This raises the research question of whether MCG may be useful for the early triage of patients with acute chest pain. In the study protocol, a clinical evaluation is defined that will assess the ability of a portable MCG instrument, using a fixed algorithm, to R/O ACS, with improved safety (i.e. << 2% false negative rate) in patients presenting to an emergency setting with chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient presents to the ED with chest pain syndrome of suspected cardiac origin (i.e. symptoms consistent with ACS)
* 18+ year old male or female
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* ST-segment Elevation MI (STEMI)
* Clear non-ischaemic cause for symptoms (e.g. trauma)
* Haemodynamic instability on admission (e.g. BP>220mmHg systolic & >110mmHg diastolic, <80mmHg systolic & <40mmHg diastolic, HR>160bpm)
* Ventricular tachycardia or fibrillation that cannot be treated effectively
* Atrial fibrillation
* Thoracic metal implants
* Pacemaker or internal defibrillator
* Pregnancy (if after 20-week period)* or lactation
* Patient unable to lie down (i.e. supine position) or stay still on the examination bed
* Patient unable to understand the informed consent process and/or has a poor understanding of English (e.g. English-speaking relative/translator not available)
* Patient unable to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that present to the ED with chest pain syndrome of suspected cardiac origin (i.e. symptoms consistent with ACS) who are in normal sinus rhythm
Sampling Method: Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of MCG | at discharge, 3 months follow-up
  Sensitivity and specificity for diagnosing ACS, focusing on rule-out, in chest pain patients with normal sinus rhythm

SECONDARY OUTCOMES:
Proportion of adverse events and types | at discharge, 3 months follow-up
All-cause mortality (divided into CV and non-CV causes) proportion | through 1 week and 3 months follow-up
Change in sensitivity and specificity for diagnosing ACS, focusing on rule-out, in chest pain patients with normal sinus rhythm, according to low, intermediate and high PTP groups | at discharge, 3 months follow-up
MACE post-presentation to the ED (rule-out of ACS divided into MCG vs reference standard [adjudicated ACS/non-ACS diagnose]) | through 1 week and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Steve Goodacre, MB ChB MRCP DiplMC FCEM, Principal Investigator — University of Sheffield; Sheffield, UK
Locations (5):
- United Kingdom (5):
  - Southmead Hospital, North Bristol NHS Trust, Bristol
  - Leicester Royal Infirmary, Univeristy Hospitals of Leicester NHS Trust, Leicester
  - St George's University Hospitals NHS Foundation Trust, London
  - Queens Medical Centre, Nottingham Univeristy Hospitals NHS Trust, Nottingham
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No